CLINICAL TRIAL: NCT04477902
Title: A Longitudinal, Long-Term, Observational Study of COVID-19 Experience and Health Effects
Brief Title: Long-Term Experience and Health Effects of COVID-19
Status: Completed | Type: Observational
Sponsor: Altura (Industry)
Responsible Party: Sponsor
Other Study IDs: altcovid-192020
Record Dates: First submitted 2020-07-16; First posted 2020-07-20 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2020-07

CONDITIONS: Covid19; Corona Virus Infection; Quality of Life; Risk Reduction
Keywords: covid-19; corona virus; covid19; coronavirus; SARS-CoV-2; infection; household; transmission; vaccine; clinical trials; online; Altura; outpatient; telemedicine
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Risk Reduction Behavior; Infections

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: none - observational — online survey

SUMMARY:
The purpose of this study is to gain on-going COVID-19 feedback/data to drive timely action locally and nationally in order to mitigate transmission. Data will be deidentified and consolidated to create a large national longitudinal database.

DETAILED DESCRIPTION:
Ths is a longitudinal, observational, descriptive study to gather data needed to support a better understanding of COVID-19 from the perspective of a diverse national population.

This multi-phase study will use an action research approach to identify specific ways that physician groups, federally qualified health centers (FQHCs), public health departments, and other health and social services systems in the United States can address healthcare needs and mitigate the transmission of COVID-19. Email surveys will be used to assess the historical and current status of participants by medical condition, geography, and demographic characteristics, as well as their history of symptoms (e.g. recent cough, fever, loss of sense of taste or smell, etc.) and their current psychosocial needs.

The study will provide the structure for an iterative exploration of trends over time (up to 24 months). The opt-in survey will be posted and available to individuals 18 and older who choose to participate. Survey frequency will be every two weeks.

To analyze broader trends, all survey responses will be de-identified and aggregated. Overall general findings will not be linked to individuals or physician groups when reporting and publishing study results.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Any gender specification
* Has consented to proceed with survey
* Is able to complete the survey via email on a regular basis

Exclusion Criteria:

* none

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Anyone in the USA can participate in this study that meets inclusion criteria. To ensure diversity urban, suburban and rural areas of the country will be included.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-06-22 (Actual); Study Completion 2021-06-22 (Actual)

PRIMARY OUTCOMES:
Longitudinal survey | 2 years
  To gain on-going COVID-19 feedback/data to drive timely action locally and nationally in order to mitigate transmission.

CONTACTS AND LOCATIONS:
Overall Officials: Pete Fronte, MBA, Study Chair — Altura
Locations (1):
- Altura, Mission Viejo, California, United States

IPD SHARING:
Plan to Share IPD: Undecided